CLINICAL TRIAL: NCT01956903
Title: Phase 1/2 Study of Treatment of Refractory Acute Graft-Versus-Host Disease After First Line Therapy by Sequential Infusion of Expanded In-Vitro Allogenic Mesenchymal Stem Cell
Brief Title: Treatment of Refractory Acute Graft-Versus-Host Disease by Sequential Infusion of Allogenic Mesenchymal Stem Cell.
Acronym: CSM/EICH2010
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de trasplantes hematopoyeticos y terapia celular (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSM/EICH2010; 2010-020947-11 (EudraCT Number)
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Graft-Versus-Host Disease
Keywords: mesenchymal stem cell transplantation
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allogenic Mesenchymal Stem Cell (Experimental): Sequential Infusion of Expanded in-Vitro Allogenic Mesenchymal Stem Cell (MSC). Dosage 0,7 x 10e6 MSC/Kg/dose (cumulative minimum dose: 2,8 x 10e6 CSM/Kg.
  Interventions: Genetic: Allogenic Mesenchymal Stem Cell

INTERVENTIONS:
Genetic: Allogenic Mesenchymal Stem Cell — Expanded in-Vitro Allogenic Mesenchymal Stem Cell (authorized by Spain, "Agencia Española de Medicamentos y Productos Sanitarios" with number 06-076)

SUMMARY:
The purpose of this study is to determine the safety and efficacy of sequential infusion of allogenic mesenchymal stem cells (MSC) expanded "in vitro" in treating patients with acute graft-versus-host disease refractory to first-line therapy.

DETAILED DESCRIPTION:
1. Ethical considerations:

   * The study will be conducted in accordance with the requirements expressed in the Declaration of Helsinki (Hong Kong revision, September 1989) and following the recommendations of the Good Clinical Practice of the Clinical Trials (document 111/3976/88, July 1990 ) and Spanish legislation (Royal Decree 561/1993, published in April 16th Official State Bulletin "BOE"; May 13th, 1993) laying down the requirements for conducting clinical drug trials.
   * Every subject will receive a written document called "Patient Information Sheet" that contains information about the following aspects of clinical trial: a) Aim of the study, methodology, study treatment and alternative therapies, expected benefits for himself or society, risks of the study and possible adverse events, number of visits and additional tests.

     b) Voluntary nature of their participation and ability to withdraw at any time, without thereby altering the doctor-patient relationship.

     c) People who have access to the data of the volunteer and how they maintain the confidentiality of the data.

     d) How to contact with the investigator if necessary.
   * The investigator will obtain the informed consent of the subject or, failing that, from a legal representative. The subject is preferably expressed written consent or, alternatively, orally to the research team independent witnesses who declare in writing under its responsibility.
   * The person participating in the clinical trial or his representative may revoke the consent at any time.
2. Data Access:

   * In order to ensure the confidentiality of the trial data, only have access to them, the researcher and his team, the test monitor and the Clinical Research Ethics Committee of the corresponding center or purposes under test and relevant health authorities.
   * Protection of data: The content of the data collection forms and the documents generated during the study, will be protected from unauthorized uses by people outside the research and, therefore, will be considered strictly confidential and will not be disclosed to third parties except to those specified in the preceding paragraph.
3. Data Collection:

   * Data colection forms will be dated and signed by the authorized principal investigator.
   * Unknown data will be collected as "NA"(not available).
   * Unusual or extreme results, or that do not match the expected sequence will be checked and corrected by initialing, signing and providing an explanation.
   * Laboratory results that exceed normal limits established by the laboratory of the center, should be checked by the researcher and their significance will be noted next to the data, by initialing and signing.
4. Statistical Analysis:

   * Baseline data will be analyzed using descriptive statistics and demographics (mean, median, standard deviation, minimum, maximum, and number of valid cases) for quantitative variables and absolute and relative frequencies for categorical variables.
   * The primary efficacy objective is to determine the response rate of graft versus host disease (confidence intervals 95%).
   * The primary safety objective is to determine the incidence of adverse events and toxicity related to the administration of the CSM (confidence intervals 95%).
   * Secondary objectives: analyze overall survival and disease-free survival by the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies who have undergone allogenic stem cell transplantation and who are diagnosed with acute graft-versus-host-disease refractory to first-line treatment.
* Patients must have adequate cardiac function without evidence of uncontrolled hypertension, congestive heart failure or myocardial infarction within 6 months prior to the process.
* Adequate pulmonary function with no evidence of severe obstructive or restrictive pulmonary disease.
* Be able to understand the information and sign the informed consent.

Exclusion Criteria:

* Patients with uncontrolled disease or in progress at the time of treatment.
* Patients with uncontrolled bacterial, viral or fungal infection.
* Patients with inadequate cardiac or pulmonary function.
* Patients who do not have the required donor.
* Women pregnant or at risk of pregnancy by inadequate contraceptive measures.
* Patients who in the opinion of the investigator are not able to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Adverse effects | from infusion to 100 days after stem cell transplant
  * Infusion related.
  * Infection Rate.

SECONDARY OUTCOMES:
efficacy | Acute Graft-Versus-Host Disease period (100 days)
  Acute Graft-Versus-Host Disease response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Fermín M Sánchez Guijo, MD, Principal Investigator — Hospital Universitario de Salamanca, Salamanca. Spain.; Felipe Prosper, MD, Principal Investigator — Clínica Universitaria de Navarra, Spain.; Eduardo Olavarría, MD, Principal Investigator — Hospital de Navarra, Spain; Rocío Parody, MD, Principal Investigator — Hospital Universitario Virgen del Rocío, Seville, Spain.; Carmen Regidor, MD, Principal Investigator — Hospital Universitario Puerta del Hierro, Spain; Carmen Martínez, MD, Principal Investigator — Hospital Clinic i Provincial de Barcelona, Spain; Rodrigo Martino, MD, Principal Investigator — Hospital de la Santa Creu i Sant Pau, Spain; José Antonio Pérez-Simón, MD, Principal Investigator — Hospital Universitario Virgen del Rocío, Seville, Spain.
Locations (1):
- Grupo Espanol de trasplantes hematopoyeticos y terapia celular, Madrid, Madrid, Spain